CLINICAL TRIAL: NCT00497523
Title: Double Blind, Multinational, Multicentre, Parallel-group, Placebo-controlled Design Trial of the Efficacy and Safety of Nebulised Beclometahsone Dipropionate (400 μg b.i.d.) Plus as Needed Salbutamol Versus as Needed Salbutamol or as Needed Salbutamol/Beclomethasone Fixed Combination, in the 12-week Treatment of Young Children With Asthma Symptoms
Brief Title: Efficacy and Safety of Nebulised Beclomethasone Dipropionate Plus as Needed Salbutamol vs as Needed Salbutamol or as Needed Salbutamol/Beclomethasone Fixed Combination in Young Children With Asthma Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC/PR/1404/002/05
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Bronchial Asthma
Keywords: Asthma; Young Children; Corticosteroids; Beclomethasone; Salbutamol; Beclomethasone/Salbutamol fixed combination; Suspension for nebulisation
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Beclomethasone dipropionate (Experimental)
  Interventions: Drug: Beclomethasone dipropionate
- Beclomethasone dipropionate/Salbutamol combination (Experimental)
  Interventions: Drug: Beclomethasone dipropionate/Salbutamol combination
- Salbutamol (Active Comparator)
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: Beclomethasone dipropionate
  Arms: Beclomethasone dipropionate
Drug: Beclomethasone dipropionate/Salbutamol combination
  Arms: Beclomethasone dipropionate/Salbutamol combination
Drug: Salbutamol
  Arms: Salbutamol

SUMMARY:
To demonstrate a superior efficacy of BDP plus rescue salbutamol suspension for nebulisation, compared to placebo plus rescue salbutamol, in the relief of symptoms of asthma in young children with persistent symptoms of asthma.

DETAILED DESCRIPTION:
Asthma is a chronic disease which is estimated to affect over 25 million people both in the US and Europe(i.e. approximately 10% of the total population).There is evidence that over the last 20 years prevalence has considerably increased, especially among children. The diagnosis of asthma in children may be difficult, largely because episodic wheezing and cough are among the common symptoms encountered in childhood illnesses, particularly in children under 3 years old.Although in these young children there is the possibility of over treatment, the episodes of wheezing may be reduced in intensity by the effective use of anti-inflammatory medications and bronchodilators rather than antibiotics. At present, pharmacological therapy is used to treat reversible airway obstruction, inflammation and hyperreactivity in both children and adults. Medications include preventive treatments in forms of antinflammatory/antiallergic agents (e.g. glucocorticosteroids, leukotriene antagonists, cromolyn sodium) and reliever treatments, in form of bronchodilators (e.g. β-adrenergic agonists, anticholinergics). Comparisons: Beclomethasone suspension for nebulisation (400 mcg U.D.V.) plus as needed salbutamol compared to placebo plus as needed salbutamol and to as needed salbutamol/beclomethasone fixed combination.

ELIGIBILITY:
Inclusion Criteria:

Patients will be enrolled into the 2-week placebo run-in period if they meet all the following criteria:

* Age ≥ 1 year and ≤ 4 years.
* At least 3 episodes of wheeze or asthma-like symptoms in the 6 months preceding the study entry.
* A cooperative attitude and ability to be trained to inhale correctly from the device and to complete the diary cards.
* Written parental/guardian informed consent obtained.

Patients will be then randomised to the treatment period if they meet all the previous criteria plus:

* Presence in at least 7 days out of the 14 days of the run-in period of at least one of the following symptoms: wheeze, cough or shortness of breath; or had required at least one dose of relief salbutamol.

Exclusion Criteria:

* History of severe asthma exacerbation or exacerbations requiring hospitalisation in the previous 4 weeks.
* Symptomatic infection of the airways requiring treatment with antibiotics or antimycotics in the previous 4 weeks.
* Treatment with inhaled steroids in the previous 4 weeks or oral steroids in the previous 8 weeks.
* Treatment with methyl-xantine derivatives in the previous 4 weeks.
* Treatment with long-acting β2-agonists in the previous 2 weeks.
* Changes in asthma medications taken on regular basis in the previous 4 weeks.
* Symptoms of asthma limited to seasonal allergen exposure.
* History of clinically significant cardiac, renal, neurologic, hepatic, endocrine or pulmonary disease (except asthma), or laboratory testing abnormalities, whose sequelae and/or treatments can interfere with the results of the present study.
* Evidence of pulmonary malformations.
* Evidence of immunological deficiency (patients to be withdrawn if diagnosed during the study).
* Cancer or any other chronic disease with prognosis < 2 years.
* Hypersensitivity to inhaled corticosteroids.
* Participation in another trial in the last 4 weeks.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 283 (Actual)
Dates: Start 2006-03; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Percentage of global (weeks 1-12) symptom-free days. | weeks 1-12

SECONDARY OUTCOMES:
Frequency and number of exacerbations (defined as a worsening of symptoms of asthma requiring extra oral or inhaled corticosteroids) | weeks 1-12
Single clinical symptoms | weeks 1-12 and every 2-week period
Nocturnal awakening due to symptoms of asthma | weeks 1-12 and every 2-week period
Use of rescue nebulised therapy | weeks 1-12 and every 2-week period
time to first exacerbation | weeks 1-12

CONTACTS AND LOCATIONS:
Overall Officials: Renato Cutrera, MD, Study Chair — Department of Pediatric Medicine, Children's Hospital and Research Institute Bambino Gesù, Rome, Italy
Locations (19):
- Poland (6):
  - Zaklad Alergologii Dzieciecej, Bialystok
  - Specjalistyczne Centrum Leczenia Dzieci i Mlodziezy, Krakow
  - Wojskovy Szpital Klinikzny, Krakow
  - Priwatna Pomoc Lekarska, Lodz
  - Alergovita, alergologia Dziecieca, Lublin
  - Priwtny Gabinet Pediatriczno - Alergologiczny, Rabka-Zdrój
- Ukraine (13):
  - City Children's Clinical Hospital n. 2, Dniepropetrovs'k State Medical Academy, Department of preliminary study of childhood disesas, Dniepropetrovsk
  - Dniepropetrovsk Regional Children's Clinical Hospital, State Medical Academy, Hospital Paediatric Department N.1, Dniepropetrovsk
  - Department of Hospital Pediatrics, Kharkiv State Medical University Region Clinical Children's Hospital n. 2, Kharkiv
  - Respiratory Diseases Children's Clinic, Institute of Phthisiology and Pulmonology,Academy of Medical Science of the Ukraine, Pulmonology, Kiev
  - Children's Hospital "OHMATDYT" Department of Pediatrics N. 1 of Kyiv Medical Academy of Postgraduate Education, Kyiv
  - Department of Clinical rehabilitation of children with bodily diseasesof Institute of Pediatrics, Obstetrics and Gynecology, Kyiv
  - Institute of Pediatrics, Obstetrics and Gynecology. Department of Children's Pulmonology Diseases and Ecological Problems of Health, Kyiv
  - Department of Paediatric and Neonatology, Odessa State Medical University, Odessa Region Clinical Children's Hospital, Odesa
  - Poltava regional children's clinical hospital, Ukranian stomatological academy, department of pediatrics, Poltava
  - Pediatrics Crimean State Medical University Pulmonology, Department of Republican Clinical Children's Hospital, Simferopol
  - Children's clinical hospital N.1, Zaporizzhya Medical Academy of post graduate education, department of pediatrics, Zaporizhya
  - City Clinical Hospital N. 1 , Zaporizzhya Medical Academy of post graduate education, department of paediatrics, Zaporizhya
  - Regional Children Clinical Hospital. Department of Pulmonology., Zaporizhya

REFERENCES:
- [Result] Papi A, Nicolini G, Baraldi E, Boner AL, Cutrera R, Rossi GA, Fabbri LM; BEclomethasone and Salbutamol Treatment (BEST) for Children Study Group. Regular vs prn nebulized treatment in wheeze preschool children. Allergy. 2009 Oct;64(10):1463-1471. doi: 10.1111/j.1398-9995.2009.02134.x. PMID 19772514
- [Result] Papi A, Nicolini G, Boner AL, Baraldi E, Cutrera R, Fabbri LM, Rossi GA. Short term efficacy of nebulized beclomethasone in mild-to-moderate wheezing episodes in pre-school children. Ital J Pediatr. 2011 Aug 22;37:39. doi: 10.1186/1824-7288-37-39. PMID 21859484